CLINICAL TRIAL: NCT01382589
Title: A Phase II Randomised Pilot Study to Compare the Efficacy and Safety of Subcutaneous, Bioresorbable Afamelanotide Implants and Narrow-Band Ultraviolet B (NB-UVB) Light in the Treatment of Nonsegmental Vitiligo
Brief Title: Afamelanotide and Narrow-Band Ultraviolet B (NB-UVB) Light in the Treatment of Nonsegmental Vitiligo
Acronym: NSV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clinuvel Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CUV101
Record Dates: First submitted 2011-06-07; First posted 2011-06-27 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-03

CONDITIONS: Vitiligo
Keywords: vitiligo; depigmentation; phototherapy; non-segmental vitiligo
MeSH Terms: conditions — Vitiligo | interventions — afamelanotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A: Afamelanotide + NB-UVB (Experimental): Subject in this arm will receive both afamelanotide implants (one implant administered every 28 days, 6 implants in total) and NB-UVB light (administered thrice weekly, 72 treatments in total)
  Interventions: Drug: Afamelanotide
- Arm B: NB-UVB alone (Active Comparator): Subjects in this arm B will receive NB-UVB light only (administered thrice weekly, 72 treatments in total)
  Interventions: Device: NB-UVB

INTERVENTIONS:
Drug: Afamelanotide — NB-UVB phototherapy with or without subcutaneous, bioresorbable Afamelanotide 16 mg implants, contained in a poly(D,L-lactide-co-glycolide) implant core released over 7-10 days following implantation
  Other Names: CUV1647
  Arms: Arm A: Afamelanotide + NB-UVB
Device: NB-UVB — NB-UVB light therapy 3-times per week, for total of 72 treatments
  Arms: Arm B: NB-UVB alone

SUMMARY:
The purpose of this study is to determine whether afamelanotide and narrow band UVB are effective in the treatment of non-segmental vitiligo (NSV).

DETAILED DESCRIPTION:
The investigational product, afamelanotide, is a synthetic analogue of the human alpha melanocyte stimulating hormone (alpha-MSH). The earliest described function of alpha-MSH is its ability to stimulate melanin synthesis in the skin and therefore stimulate pigmentation. Vitiligo is the most common depigmentation disorder. Interventions in the treatment of vitiligo include phototherapy with narrow-band (NB) ultraviolet B (UVB) irradiation (NB-UVB).

The purpose of this study is to look at the efficacy of afamelanotide, when combined with narrow-band ultraviolet B (NB-UVB) light, in patients with nonsegmental vitiligo. Afamelanotide is expected to speed up the repigmentation induced by NB-UVB light, leading to reducing frequency and doses of NB-UVB.

ELIGIBILITY:
Inclusion criteria:

* Male and female subjects with a confirmed diagnosis of nonsegmental vitiligo with 15% to 50% of total body surface involvement
* Stable or slowly progressive vitiligo over a 3-month period
* Aged 18 or more
* Fitzpatrick skin types III-VI
* Willing and able to comply with the conditions specified in this protocol and study procedures in the opinion of the Investigator
* Providing written Informed Consent prior to the performance of any study-specific procedure

Exclusion criteria:

* Fitzpatrick skin types I-II
* Vitiligo involving the hands and feet only
* Extensive leukotrichia, in the opinion of the Investigator
* Vitiligo of more than 5 years duration
* Allergy to afamelanotide or the polymer contained in the implant or to lignocaine/lidocaine or other local anaesthetic to be used during the administration of the implant
* Previous treatment with topical immunomodulators (corticosteroids, calcineurin inhibitors) for vitiligo within 4 weeks prior to the Screening Visit
* History of photosensitivity disorders
* Claustrophobia
* History of photosensitive lupus
* Any active and/or unstable autoimmune disease judged to be clinically significant by the Investigator
* History of melanoma or lentigo maligna
* History of dysplastic nevus syndrome
* Any malignant skin lesions
* Any skin disease that may interfere with the study evaluation
* Any evidence of organ dysfunction or deviation from normal in clinical or laboratory determinations judged to be clinically significant by the Investigator
* History of systemic or psychiatric disease judged to be clinically significant by the Investigator and which may interfere with the study evaluation
* Female who is pregnant (confirmed by positive β-HCG pregnancy test) or lactating
* Female of child-bearing potential (pre-menopausal, not surgically sterile) not using adequate contraceptive measures (i.e. oral contraceptives, diaphragm plus spermicide, intrauterine device) during the trial and for a period of three months thereafter
* Sexually active man with a partner of child-bearing potential not using barrier contraception during the trial and for a period of three months hereafter
* Participation in a clinical trial for an investigational agent within 30 days prior to the Screening Visit
* Use of any prior and concomitant therapy which may interfere with the objective of the study, including drugs that cause photosensitivity or skin pigmentation within 60 days prior to the Screening Visit
* Subjects assessed as not suitable for the study in the opinion of the Investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-09; Primary Completion 2012-07 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To compare the efficacy of afamelanotide implants and NB-UVB light in the treatment of nonsegmental vitiligo | 6 months
  Time to onset of repigmentation of full body, face, trunk and extremities Pigmentation by VASI and VETF Maintenance of pigmentation Dermatology Life Quality Index (DLQI)
  Safety of the treatment will be assessed by:
  For selected study sites, immunomodulatory assessment Full body anterior and posterior photography Vitiligo lesion photography Examination of the skin and oral mucosa and digital photography Ophthalmologic examination

SECONDARY OUTCOMES:
Maintenance of pigmentation achieved | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Leone, MD, Principal Investigator — San Gallicano Dermatological Institute, Photodermatology Unit, Roma, ITALY